CLINICAL TRIAL: NCT00313781
Title: A Phase 2, Randomized, Non-Comparative, Two-Arm Open Label, Multiple-Center Study Of CP-751,871 In Combination With Docetaxel/Prednisone In Chemotherapy- Naive (Arm A) And Docetaxel/Prednisone Refractory (Arm B) Patients With Hormone Insensitive Prostate Cancer
Brief Title: Study of CP-751,871 in Combination With Docetaxel and Prednisone in Patients With Hormone Insensitive Prostate Cancer (HRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021011
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-03

CONDITIONS: Prostatic Neoplasms
Keywords: randomized; non-comparative; efficacy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — figitumumab; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): For patients treated with docetaxel and prednisone only, who progress during treatment, CP-751,871 will be added to the regimen to test reversibility of chemoresistance.
  Interventions: Drug: CP-751,871; Drug: docetaxel; Drug: prednisone
- B (Active Comparator)
  Interventions: Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: CP-751,871 — CP-750,871 is administered intravenously at a dose of 20 mg/kg on day 1 of each 21-day cycle (for patient convenience and logistical management, the dose of CP-751,871 may be deferred up to 7 days).
  Arms: A
Drug: docetaxel — Docetaxel is administered IV on day 1 of each 21-day cycle, at a dose of 75 mg/m2.
  Arms: A
Drug: prednisone — Prednisone is administered at a dose of 5 mg twice daily.
  Arms: A
Drug: docetaxel — Docetaxel is administered IV on day 1 of each 21-day cycle, at a dose of 75 mg/m2.
  Arms: B
Drug: prednisone — Prednisone is administered at a dose of 5 mg twice daily.
  Arms: B

SUMMARY:
To test the efficacy of CP-751,871 combined with docetaxel and prednisone in the treatment of prostate cancer that is refractory to hormone therapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic, progressive hormone refractory prostate cancer
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

* Previous treatment with chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2006-05; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (5):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Orange, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
- Pfizer Investigational Site, Montreal, Quebec, Canada
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, München
- Spain (3):
  - Pfizer Investigational Site, A Coruña, A Coruña
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
- Pfizer Investigational Site, Sankt Gallen, Switzerland
- United Kingdom (3):
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Guildford

REFERENCES:
- [Derived] de Bono JS, Piulats JM, Pandha HS, Petrylak DP, Saad F, Aparicio LM, Sandhu SK, Fong P, Gillessen S, Hudes GR, Wang T, Scranton J, Pollak MN. Phase II randomized study of figitumumab plus docetaxel and docetaxel alone with crossover for metastatic castration-resistant prostate cancer. Clin Cancer Res. 2014 Apr 1;20(7):1925-34. doi: 10.1158/1078-0432.CCR-13-1869. Epub 2014 Feb 17. PMID 24536060
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021011&StudyName=Study%20of%20CP-751%2C871%20in%20Combination%20With%20Docetaxel%20and%20Prednisone%20in%20Patients%20with%20Hormone%20Insensitive%20Prostate%20Cancer%20%28HRPC%29

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-751,871+Docetaxel+Prednisone: Participants received docetaxel 75 milligram(mg)/square meter(m^2) infusion intravenously (IV) over 1 hour on Day 1, followed by CP-751,871 20 mg/kilogram (kg) infusion IV on Day 1 along with prednisone 5 mg twice daily (BID) in a 21 days cycle, up to 17 cycles.
- Docetaxel+Prednisone: Participants received docetaxel 75 mg/m^2 infusion IV over 1 hour on Day 1 along with prednisone 5 mg BID in a 21 days cycle, up to 17 cycles.
- Docetaxel+Prednisone+CP-751,871 Crossover: Participants from the "Docetaxel+Prednisone" group who, after disease progression while receiving docetaxel and prednisone alone, opted to receive CP-751,871 20 mg/kg infusion IV on Day 1 of a 21 days cycle, along with docetaxel 75 mg/m^2 infusion IV over 1 hour on Day 1 and prednisone 5 mg BID, up to 17 cycles.
Period: Before Crossover
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Started | 102 | 102 | 0
Treated | 97 | 102 | 0
Completed | 27 | 23 | 0
Not Completed | 75 | 79 | 0
Not completed — Death | 22 | 8 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Other | 45 | 30 | 0
Not completed — Crossover | 0 | 37 | 0
Not completed — Randomized, not treated | 5 | 0 | 0
Period: After Crossover
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Started | 0 | 0 | 37
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 27
Not completed — Death | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Other | 0 | 0 | 18

BASELINE CHARACTERISTICS:
Groups:
- CP-751,871+Docetaxel+Prednisone: Participants received docetaxel 75 milligram(mg)/square meter(m^2) infusion IV over 1 hour on Day 1, followed by CP-751,871 20 mg/kilogram (kg) infusion IV on Day 1 along with prednisone 5 mg twice daily (BID) in a 21-days cycle, up to 17 cycles.
- Total: Total of all reporting groups
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Customized [Number; unit: Participants]
  Less than (<) 18 years | 0 | 0 | 0
  18 to 44 years | 0 | 1 | 1
  45 to 64 years | 26 | 32 | 58
  Greater than or equal to (>=) 65 years | 76 | 69 | 145
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 102 | 102 | 204

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Best Response
Description: Percentage of participants with PSA best response of either PSA normalization (PN) or partial PSA response (PR) relative to the total number of participants evaluable for response. PN was defined as PSA =< 0.2 nanogram/milliliter (ng/ml) on 2 successive evaluations at least 3 weeks apart and no imaging or clinical evidence of disease progression. PP was defined as >= 50% decrease in PSA from baseline on 2 successive evaluations at least 3 weeks apart and no imaging or clinical evidence of disease progression.
Time Frame: Baseline, Day 1 and Day 15 of each cycle, end of treatment (up to 28 days post last dose) and follow-up (monthly, up to 150 days post last dose)
Population: Response-evaluable population: All enrolled participants who had a baseline PSA reference value and received at least one dose of assigned treatment with the exception of those participants without symptomatic or objective progression (participants with PSA progression only) who withdraw consent prior to Cycle 3.
Measure: Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 87 | 98 | 32
Percentage of participants | 51.7 [42.4 to 61.0] | 60.2 [51.4 to 68.5] | 28.1 [15.5 to 43.9]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to first event of disease progression. Disease progression events were defined as the following: PSA progression,objective disease progression as per RECIST, death, and discontinuation of treatment due to symptomatic deterioration. PSA progression was defined as the time-point of PSA progression on 2 successive evaluations taken 1 week apart after dosing in cycle 3.
Time Frame: Baseline, Day 15 of each cycle and follow-up (monthly, up to 150 days post last dose)
Population: Full analysis set included all participants who were enrolled into the study and received at least one assigned treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 97 | 102 | 37
Months | 4.9 [4.1 to 5.9] | 7.7 [6.1 to 8.9] | 4.0 [3.3 to 4.8]

3. Secondary Outcome: Human Anti-human Antibody (HAHA) at Baseline (Day 1 of Cycle 1)
Description: Levels of HAHA in serum were detected at baseline.
Time Frame: Baseline (Day 1 of Cycle 1)
Population: All participants who were enrolled in the study, received at least one assigned treatment and had available HAHA assessment.
Measure: Mean (Standard Deviation); unit: mg/deciliter (dl)
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone
Number analyzed (Participants) | 49 | 41
mg/deciliter (dl) | 1130.3 (406.49) | 1338.1 (804.30)

4. Secondary Outcome: Human Anti-human Antibody (HAHA) at the Last Follow-up Visit
Description: Levels of HAHA in serum were detected at the last follow-up visit.
Time Frame: The last follow-up visit (150 days post last dose)
Population: All participants who were enrolled in the study, received at least one assigned treatment and had HAHA available assessment.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 32 | 13 | 14
mg/dl | 944.81 (946.42) | 819.00 (487.94) | 970.86 (295.28)

5. Secondary Outcome: Population PK Parameters of CP-751,871
Description: Population pharmacokinetic analysis involved mixed effects modeling using nonlinear mixed effects modeling (NONMEM) software. The intent of this analysis was to establish a basic population pharmacokinetic model for CP-751,871 and to determine inter-individual and residual variability in population clearance, and volume of distribution of drug. Relationship of demographic variables (gender, age, body weight, height and ethnicity), concomitant medications and measures of altered hepatic and renal function were examined by fitting measured CP-751,871 concentrations
Time Frame: Days 1, 8 and 15 of each cycle and last follow-up visit (150 days post last dose)
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: ng/mL

6. Secondary Outcome: Total Number of Circulation Tumor Cells (CTCs)
Description: Blood samples were collected and processed to enumerate the number of total CTCs via Veridex CellSearch technology in which CTCs were identified based on cell surface positive epithelial cell adhesion molecule (EpCAM) and cytokeratin staining.
Time Frame: Baseline, prior to dosing in odd numbered cycles (ie. Cycle 1, 3, 5, etc) and end of treatment (up to 28 days post last dose)
Population: Participants who were enrolled to the study were included in the analysis. n = number of participants with evaluable data at each timeframe.
Measure: Mean (Standard Deviation); unit: Number of CTCs/7.5 mL
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone
Number analyzed (Participants) | 46 | 39
Number of CTCs/7.5 mL
  Baseline (Cycle 1 Day 1) (n=46, 39) | 105.17 (259.60) | 213.23 (555.82)
  Cycle 3 Day1 (n=28, 29) | 6.39 (11.39) | 12.21 (27.52)
  Cycle 5 Day 1 (n=25, 23) | 15.20 (46.40) | 17.78 (28.11)

7. Secondary Outcome: Total Number of the Insulin Like Growth Factor Receptor Type 1 (IGF-1R) Positive CTCs
Description: Blood samples were collected to enumerate the number of total IGF-1R positive CTCs via Veridex CellSearch technology in which CTCs were identified based on cell surface positive EpCAM and cytokeratin staining. A separate CellSave tube of cells was also collected and processed with cell surface staining of IGF-1R to enumerate surfaces of IGF-1R-positive CTCs.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Number of IGF-1R positive CTCs/7.5 mL
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone
Number analyzed (Participants) | 22 | 18
Number of IGF-1R positive CTCs/7.5 mL
  Baseline (Cycle 1 Day 1) (n=22, 18) | 24.73 (25.32) | 54.94 (55.52)
  Cycle 3 Day1 (n=12, 15) | 2.33 (4.48) | 4.93 (7.74)
  Cycle 5 Day 1 (n=11, 10) | 2.00 (4.49) | 3.90 (6.03)

8. Secondary Outcome: Quality of Life Measured by the Functional Assessment of Cancer Treatment-Prostate (FACT-P)
Description: The FACT-P was a 39-item participant questionnaire which assesses physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and additional prostate cancer specific concerns (12 items). All items were scored from 0 (not at all) to 4 (very much). The total FACT-P score ranged from 0-156, with higher scores representing a better QoL with fewer symptoms. A score of 156 represented the best outcome.
Time Frame: Baseline, Cycle 1 to Cycle 10 before drug administration and end of treatment (up to 28 days post last dose)
Population: The summary table was not provided based on 1) the negative primary finding of the study that CP-751,871 did not improve response in CP-751,871+Docetaxel + Prednisone and had significantly worse PFS than Docetaxel +Prednisone, which rendered the patient reported outcome (PRO) summary irrelevant 2) lack of resources as the program was terminated.
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Pain Measured by the Modified Brief Pain Inventory-Short Form (mBPI-sf Modified Pfizer)
Description: The mBPI-sf was a self administered questionnaire developed to assess pain severity and pain interference with functional activities during a 24-hour period prior to evaluation. For the worst pain item of the mBPI-sf scale (11 point Likert scale; range: 0 [no pain] to 10 [pain as bad as you can imagine]), participants were asked to rate their pain by marking an "X" in one of the 10 boxes that best described their pain at its worst in the last 24 hours post surgery and at least 12 hours after discontinuation of the peripheral nerve block or neuraxial block.
Time Frame: Baseline, Cycle 1 to Cycle 10 before drug administration and end of treatment (up to 28 days post last dose)
Population: The summary table was not provided based on 1) the negative primary finding of the study that CP-751,871 did not improve response in CP-751,871+Docetaxel + Prednisone and had significantly worse PFS than Docetaxel +Prednisone, which rendered the PRO summary irrelevant 2) lack of resources as the program was terminated.
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) for CP-751,871
Description: Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration.
Time Frame: Days 1, 8 and 15 of each cycle and last follow-up visit (150 days post last dose)
Population: The summary table of this outcome measure was not provided based on lack of resources as the program was terminated.
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for CP-751,871
Time Frame: Days 1, 8 and 15 of each cycle and last follow-up visit (150 days post last dose)
Population: The summary table of this outcome measure was not provided based on lack of resources as the program was terminated.
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for CP-751,871
Time Frame: Days 1, 8 and 15 of each cycle and last follow-up visit (150 days post last dose)
Population: The summary table of this outcome measure was not provided based on lack of resources as the program was terminated.
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUC0-tau) for CP-751,871
Time Frame: Days 1, 8 and 15 of each cycle and last follow-up visit (150 days post last dose)
Population: The summary table of this outcome measure was not provided based on lack of resources as the program was terminated.
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. 199 out of 204 participants were treated.
Arm/Group | CP-751,871+Docetaxel+Prednisone | Docetaxel+Prednisone | Docetaxel+Prednisone+CP-751,871 Crossover
Serious Adverse Events (participants affected / at risk) | 64/97 | 37/102 | 20/37
Other Adverse Events (participants affected / at risk) | 96/97 | 53/102 | 21/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871+Docetaxel+Prednisone (N=97) | Docetaxel+Prednisone (N=102) | Docetaxel+Prednisone+CP-751,871 Crossover (N=37)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 7 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1
Asthenia (General disorders) | 4 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Death (General disorders) | 2 | 0 | 0
Disease progression (General disorders) | 8 | 3 | 6
Drug interaction (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 0 | 3
Pyrexia (General disorders) | 1 | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 4 | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 3 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 4 | 2
Salmonellosis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Bladder tamponade (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871+Docetaxel+Prednisone (N=97) | Docetaxel+Prednisone (N=102) | Docetaxel+Prednisone+CP-751,871 Crossover (N=37)
Anaemia (Blood and lymphatic system disorders) | 13 | 21 | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 22 | 24 | 4
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 8 | 10 | 4
Neutropenia (Blood and lymphatic system disorders) | 34 | 37 | 10
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 7 | 1 | 1
Deafness bilateral (Ear and labyrinth disorders) | 2 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 6 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 7 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 2 | 3 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 1
Conjunctival pallor (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 6 | 5 | 2
Dry eye (Eye disorders) | 2 | 0 | 0
Ectropion (Eye disorders) | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 2 | 0
Eye pain (Eye disorders) | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0
Keratoconjunctivitis sicca (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 9 | 8 | 6
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0
Scleral haemorrhage (Eye disorders) | 2 | 0 | 0
Vision blurred (Eye disorders) | 5 | 5 | 2
Visual impairment (Eye disorders) | 0 | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 5 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Anal inflammation (Gastrointestinal disorders) | 3 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 22 | 17 | 8
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 64 | 38 | 14
Dry mouth (Gastrointestinal disorders) | 6 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 8 | 6 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 2
Faecal incontinence (Gastrointestinal disorders) | 2 | 2 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 2
Frequent bowel movements (Gastrointestinal disorders) | 1 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 3 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 5 | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 1 | 1 | 2
Gingivitis (Gastrointestinal disorders) | 2 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 5 | 3 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 34 | 28 | 10
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 4 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 5 | 2 | 3
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 10 | 6 | 2
Rectal tenesmus (Gastrointestinal disorders) | 4 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 1 | 0
Steatorrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 18 | 8 | 3
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 19 | 12 | 10
Vomiting projectile (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 38 | 33 | 13
Catheter site pruritus (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 4 | 1
Chest pain (General disorders) | 2 | 3 | 2
Chills (General disorders) | 6 | 6 | 3
Death (General disorders) | 0 | 0 | 1
Device occlusion (General disorders) | 0 | 1 | 0
Discomfort (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1
Energy increased (General disorders) | 0 | 1 | 0
Extravasation (General disorders) | 1 | 2 | 0
Face oedema (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 40 | 36 | 14
Feeling cold (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 1 | 0
Gait disturbance (General disorders) | 2 | 2 | 2
General physical health deterioration (General disorders) | 2 | 0 | 2
Influenza like illness (General disorders) | 0 | 1 | 1
Infusion site pruritus (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 1 | 0
Irritability (General disorders) | 2 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 3 | 0
Mucosal dryness (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 15 | 12 | 1
Oedema (General disorders) | 1 | 2 | 2
Oedema peripheral (General disorders) | 10 | 28 | 4
Pain (General disorders) | 6 | 3 | 4
Premature ageing (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 12 | 13 | 4
Sensation of pressure (General disorders) | 0 | 1 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0
Therapeutic response unexpected (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Ulcer (General disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0 | 1
Allergic oedema (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 1
Candidiasis (Infections and infestations) | 2 | 3 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 1 | 0
Gastric infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Genital candidiasis (Infections and infestations) | 1 | 0 | 0
Gingival infection (Infections and infestations) | 3 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 3 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0
Localised infection (Infections and infestations) | 3 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 4 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 4 | 0
Nasopharyngitis (Infections and infestations) | 7 | 11 | 4
Onychomycosis (Infections and infestations) | 2 | 5 | 2
Oral candidiasis (Infections and infestations) | 4 | 4 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Oral viral infection (Infections and infestations) | 0 | 1 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 2 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 4 | 3 | 2
Rhinitis (Infections and infestations) | 3 | 6 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 2 | 0
Tooth infection (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 0
Urinary tract infection (Infections and infestations) | 12 | 7 | 2
Viral infection (Infections and infestations) | 1 | 1 | 0
Wound infection (Infections and infestations) | 2 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chemical injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 4 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Alanine aminotransferase (Investigations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 1 | 0
Aspartate aminotransferase (Investigations) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase (Investigations) | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 4 | 3
Blood amylase increased (Investigations) | 2 | 2 | 1
Blood bicarbonate decreased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 2 | 1
Blood creatinine increased (Investigations) | 9 | 0 | 2
Blood glucose (Investigations) | 1 | 0 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 4 | 3 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0
Blood magnesium increased (Investigations) | 0 | 1 | 0
Blood phosphorus (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 1 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 2 | 1
Blood urea increased (Investigations) | 4 | 1 | 2
Blood uric acid increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 3 | 1
General physical condition abnormal (Investigations) | 0 | 1 | 1
Granulocyte count decreased (Investigations) | 0 | 1 | 0
Haemoglobin (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 2 | 1
International normalised ratio abnormal (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Lymphocyte count (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Murphy's sign positive (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 2 | 0
Neutrophil count increased (Investigations) | 1 | 1 | 0
Platelet count (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 2 | 2 | 1
Platelet count increased (Investigations) | 0 | 1 | 0
Renal function test abnormal (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 1 | 0
Weight decreased (Investigations) | 18 | 8 | 6
Weight increased (Investigations) | 1 | 3 | 1
White blood cell count (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 4 | 3 | 0
White blood cell count increased (Investigations) | 2 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Central obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 56 | 32 | 20
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 34 | 15 | 14
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 4 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 4 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 13 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Joint stiffness (Metabolism and nutrition disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 7 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 | 11 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 8 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 13 | 4
Myopathy (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 18 | 10
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ageusia (Nervous system disorders) | 2 | 3 | 1
Amnesia (Nervous system disorders) | 5 | 1 | 2
Aphonia (Nervous system disorders) | 2 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 4 | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 10 | 16 | 6
Dizziness exertional (Nervous system disorders) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Drooling (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 37 | 37 | 12
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 9 | 7 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 8 | 2
Hypogeusia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 15 | 16 | 5
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 3 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 16 | 22 | 12
Neurotoxicity (Nervous system disorders) | 9 | 3 | 0
Paraesthesia (Nervous system disorders) | 7 | 15 | 5
Paraparesis (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 5 | 4
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 2 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 0
Sleep phase rhythm disturbance (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 1
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 2 | 4 | 1
Tremor (Nervous system disorders) | 6 | 2 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 7 | 2 | 1
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 4 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 3 | 3 | 1
Depression (Psychiatric disorders) | 7 | 1 | 2
Disorientation (Psychiatric disorders) | 8 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 12 | 1
Listless (Psychiatric disorders) | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 1 | 1
Nervousness (Psychiatric disorders) | 1 | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 5 | 3 | 2
Enuresis (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 7 | 3 | 3
Haemoglobinuria (Renal and urinary disorders) | 1 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 1
Incontinence (Renal and urinary disorders) | 2 | 1 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 8 | 9 | 4
Pollakiuria (Renal and urinary disorders) | 5 | 4 | 2
Polyuria (Renal and urinary disorders) | 4 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 3 | 3
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 7 | 4 | 3
Urinary retention (Renal and urinary disorders) | 7 | 2 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 1
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 2
Gynaecomastia (Reproductive system and breast disorders) | 0 | 2 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 4 | 3
Penile pain (Reproductive system and breast disorders) | 1 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 2 | 1
Prostatic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 13 | 5
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 23 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 15 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 46 | 51 | 17
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 14 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 8 | 10 | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hair disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 7 | 15 | 7
Nail toxicity (Skin and subcutaneous tissue disorders) | 6 | 6 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 4 | 6 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4 | 2
Purpura (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 9 | 7 | 2
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin fragility (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Skin toxicity (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 4
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Denture wearer (Social circumstances) | 1 | 0 | 0
Capillary fragility (Vascular disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2 | 1
Flushing (Vascular disorders) | 3 | 8 | 1
Haematoma (Vascular disorders) | 5 | 2 | 1
Hot flush (Vascular disorders) | 1 | 6 | 0
Hypertension (Vascular disorders) | 3 | 4 | 2
Hypotension (Vascular disorders) | 8 | 5 | 1
Intermittent claudication (Surgical and medical procedures) | 1 | 1 | 0
Intra-abdominal haematoma (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Pallor (Vascular disorders) | 8 | 1 | 3
Peripheral embolism (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.